CLINICAL TRIAL: NCT04807452
Title: Effects of Strength And Balance Training on Diabetic Peripheral Neuropathy
Brief Title: Strength And Balance Training on Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00667 Farhan Haleem
Record Dates: First submitted 2020-12-21; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Resistance Training; Diabetic Neuropathies; Quality of Life; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength and balance training (Active Comparator): Exercises like ROMS, stretching, static balance and dynamic balance
  Interventions: Other: Strength and balance training
- Aerobics training (Experimental): Control Group received aerobic training.
  Interventions: Other: Aerobics training

INTERVENTIONS:
Other: Strength and balance training — Passive ROM to possible level of knee (flexion and extension), ankle (dorsiflexion and plantar flexion), forefoot (inversion and eversion) and toe (flexion and extension, adduction and abduction) joints.Resisted flexion and extension of knee, dorsiflexion and planter flexion of ankle, inversion and eversion of foot, flexion/extension, and abduction/adduction of toe with help of thera-band.The exercise prescription for strength training was made at approximately 50% of the estimated 1-RM. Exercise progression was achieved by instructing participants to increase the weight lifted in a specific exercise when they could perform 2 sets of 10-12 repetitions without maximal exertion on 2 consecutive training days. On basis of Borg Rating of Perceived Exertion of 10 to 13.Tandem leg stance for first 2 weeks and then it was progressed to Single leg stance toe and heel stance.For dynamic balance:backward walk Tandem walk and sideways walk.
  Arms: Strength and balance training
Other: Aerobics training — After the baseline assessment, the participant in the Group B received Aerobic exercise with routine medical care.
  All patients were followed for 3 days a week for 8 weeks treatment. Control Group received aerobic training. Control group received stretching exercise for 10 minutes and then treadmill walk for 10 minutes and then stationary bicycle for 10 minutes, and steppers for 10 minutes and 5 minute cool down .
  Arms: Aerobics training

SUMMARY:
A Randomized Control Trial was conducted on 20 participants, equally allocated in strength plus balance and aerobic group from February-2020 until December-2020.Participants were selected according to inclusion and exclusion criteria on purposive sampling technique and randomization was done by sealed envelope method. Inclusion criteria was both gender, 40 years to 80 years, Patients with type 2 diabetes ,diabetic peripheral neuropathy and Toronto neuropathy score 6 or greater. Participants were assessed after taking consent before and after 12 sessions through Toronto clinically neuropathy system, SF-36 and berg balance scale. Data was analyzed using SPSS v.22.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) adds to decrease functional performance in people with diabetes. People having DPN found to have decrease proprioception, decrease muscle strength specifically in dorsiflexion and planter-flexors of foot and decrease ankle mobility. An important result of DPN on skeletal muscle is speeded motor axon loss. The injuries to motor units have been found in intrinsic foot and hands muscles as well as dorsiflexion of lower limb. Declined muscle strength with DPN has been told in a number of muscles, counting plantar flexor and dorsi-flexors of ankle, flexor and extensor of knee. As predicted, the peripheral ankle muscles have more decline in strength as compared thigh muscle. M.Davies stated in his study that DPN has a negative effect on the quality of life of an individual.In "Painful diabetic peripheral neuropathy", the emotional and physical of quality of life are markedly changed, and associated anxiety, sleep disturbance and depression are found in 43% of the affected population. Occupation status in 35 to 43% of patients were affected, within job patients, as a result of pain, admit an usual of 5.5 missed workdays/month (30). Besides compromised life quality, patients with DPN also have greater fall risk due to imbalance problem and this risk is probable high in older age, associated depression and severity of DPN. Consequently, falls and broken bones are common among patients affected, occurring in around 25% of adults greater than 65 years with diabetes compared with 18% same population with no diabetes. The most common complication linked with DPN is frequent foot infections, ulcers and amputations, and Charcot's-joints. It was calculated that 15% of diabetic patients will progress to at least one foot ulcer, and one latest study witnessed a yearly occurrence of approximately 2%. It has been stated that 60%-70% of foot ulcers caused by diabetes are neuropathic in nature .Worldwide incidence of foot ulcer is 6.3%, and the occurrence in Africa, North America, Europe, Oceania and Asia was 7.2%, 13.0%, and 5.1%, 3.0% and 5.5% respectively. A literature also described the occurrence of diabetic foot in Pakistan around 7.6%, with more prevalent in men than women. Other difficulties of DPN contains imbalance, greater fall risk, psychosocial problems, mobility restriction, and sever case can lead to amputation thus restricting patient socially and has severely negative effect on patients life.There is very little data available on the effects of DPN on mortality.Elder individuals have a greater frequency of neuropathy than younger people, and are 17 times more likely to fall. It is crucially important to improve strength and in patients having large nerve fiber involvement. Elder can take benefit from intense strength training by improving coordination, increasing muscle strength and balance, and thus dropping fall and fracture risk. Resistance exercise is suggested for patients having diabetes type 2 and controlling mass of skeletal muscle (sarcopenia) with high resistance (1 RM) 2 to 4 days/week. Both side ankle ROM exercise, functional balance exercises like sit to stand, gait training for reduction planter load , Proprioceptive training exercise such as, stepping with alternate feet, balance board training (prevention of fall) .Several studies were also carried on effects of aerobic exercises and reported quit good effects. A literature review was done in the year 2019. Study concluded that among different physical therapy approaches, Aerobic exercise is best for reducing diabetic risk factors including diabetic neuropathy. In the year 2017, S.Billinger conducted a trail on aerobic exercises. Objectives of the study were to find the effects of aerobic exercises on vascular health. Duration of the study was 16 weeks and study reported that there is slight improvement in the vascular health of diabetic patients. Further 2 trails were conducted by S.Dixit in the year 2013 and 2014. Main objective of the study was to evaluate the effects of aerobic exercise on quality of life and progression of diabetic neuropathy respectively. Study stated the positive effects of aerobic training that I could improve the quality of life and slow down the progression of DPN.Another study was done by A.Waje in the year 2020. Study was based on the comparison of balance training exercise with PNF and its effects on balance. Study reported positive effects of both exercises but also report great effects when both treatments were given combined. K.Venkataraman et al conducted a study on short term effects of strength and balance training on functional status and quality of life in patients with diabetic neuropathy. Study claimed that strength and balance training can improve functional status, but failed to report its effects on quality of life and severity of diabetic neuropathy.Different studies were done on effects of PNF on balance and functional status in DPN. A study was done by K.Singh in the year 2016 on the effects of Proprioceptive Neuromuscular Facilitation (PNF) therapy in improving sensorimotor functions. Study claimed that PNF approach can improve the sensorimotor functions of diabetic neuropathic patients .Regarding Proprioceptive treatment, a study was done in the year 2012 by A.El-Wishy. Study was carried out in Egypt on 28 individuals. Purpose of the research was to know and equate the effects of proprioceptive exercises and conventional exercises on balance. Study reported that combination of proprioceptive and conventional exercises were more effective than isolated conventional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes (diagnosed by physician)
* Patients with diabetic peripheral neuropathy (diagnosed by Diabetic neuropathy symptom score)
* Age limit 40 to 80 years
* Patients having Toronto neuropathy score 6 or greater

Exclusion Criteria:

* Patients having ulceration/infection of feet
* Medical/Surgical conditions limiting functional mobility
* Non-ambulatory patients
* Who are not willing to participate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Toronto Clinical Neuropathy Scoring System | 4th week
  This tool is used for assessing changes from baseline. This is a quantitative scoring system for evaluating the severity of peripheral neuropathy primarily for the feet. Total score ranges from normal=0 to maximum= 19.
  Interpretation:
  * No neuropathy 0-5 points
  * Mild neuropathy 6-8 points
  * Moderate neuropathy 9-11 points
  * Severe neuropathy 12+ points Toronto Clinical Neuropathy Scoring System has good inter-class reliability (Cronbach's alpha 0.86). It is a valid instrument to reflect the presence and severity of DSP as measured by sural nerve morphology and electrophysiology findings, and morphological changes in DSP. This evidence suggests that the Toronto CSS may prove useful in documenting and monitoring DSP in the clinic and in clinical research trials.

OTHER OUTCOMES:
Health Related Quality of Life Short Form 36 v2 | 4th week
  his tool is used for assessing changes from baseline. The Short Form 36 (SF-36) was standardized in 1990 as a self-report measure of functional health and well-being. The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items) (57).Most of studies examined the reliability of the SF-36 have exceeded 0.80.Total score ranges from0-100, the lower the score, t Estimates of reliability in the physical and mental sections are typically above 0.90
Berg Balance Scale | 4th week
  This tool is used for assessing changes from baseline. 14-item scale designed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. Berg balance have high validity and reliability of 0.98.
  Interpretation:
  41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang XF, Tan BK. Effects of an ethanolic extract of Gynura procumbens on serum glucose, cholesterol and triglyceride levels in normal and streptozotocin-induced diabetic rats. Singapore Med J. 2000 Jan;41(1):9-13. PMID 10783673
- [Background] Venkataraman K, Tai BC, Khoo EYH, Tavintharan S, Chandran K, Hwang SW, Phua MSLA, Wee HL, Koh GCH, Tai ES. Short-term strength and balance training does not improve quality of life but improves functional status in individuals with diabetic peripheral neuropathy: a randomised controlled trial. Diabetologia. 2019 Dec;62(12):2200-2210. doi: 10.1007/s00125-019-04979-7. Epub 2019 Aug 29. PMID 31468106
- [Background] Davies M, Brophy S, Williams R, Taylor A. The prevalence, severity, and impact of painful diabetic peripheral neuropathy in type 2 diabetes. Diabetes Care. 2006 Jul;29(7):1518-22. doi: 10.2337/dc05-2228. PMID 16801572
- [Background] Donoghue D; Physiotherapy Research and Older People (PROP) group; Stokes EK. How much change is true change? The minimum detectable change of the Berg Balance Scale in elderly people. J Rehabil Med. 2009 Apr;41(5):343-6. doi: 10.2340/16501977-0337. PMID 19363567
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Rojhani-Shirazi Z, Barzintaj F, Salimifard MR. Comparison the effects of two types of therapeutic exercises Frenkele vs. Swiss ball on the clinical balance measures in patients with type II diabetic neuropathy. Diabetes Metab Syndr. 2017 Nov;11 Suppl 1:S29-S32. doi: 10.1016/j.dsx.2016.08.020. Epub 2016 Sep 15. PMID 27720359
- [Background] Dixit S, Maiya AG, Shastry BA. Effect of aerobic exercise on peripheral nerve functions of population with diabetic peripheral neuropathy in type 2 diabetes: a single blind, parallel group randomized controlled trial. J Diabetes Complications. 2014 May-Jun;28(3):332-9. doi: 10.1016/j.jdiacomp.2013.12.006. Epub 2013 Dec 27. PMID 24507164
- [Background] Billinger SA, Sisante JV, Alqahtani AS, Pasnoor M, Kluding PM. Aerobic exercise improves measures of vascular health in diabetic peripheral neuropathy. Int J Neurosci. 2017 Jan;127(1):80-85. doi: 10.3109/00207454.2016.1144056. Epub 2016 Feb 16. PMID 26785723
- [Background] Yaribeygi H, Butler AE, Sahebkar A. Aerobic exercise can modulate the underlying mechanisms involved in the development of diabetic complications. J Cell Physiol. 2019 Aug;234(8):12508-12515. doi: 10.1002/jcp.28110. Epub 2019 Jan 8. PMID 30623433
- [Background] Nomura T, Kawae T, Kataoka H, Ikeda Y. Assessment of lower extremity muscle mass, muscle strength, and exercise therapy in elderly patients with diabetes mellitus. Environ Health Prev Med. 2018 May 17;23(1):20. doi: 10.1186/s12199-018-0710-7. PMID 29776338